CLINICAL TRIAL: NCT07388329
Title: The Effect of Post-Scenario Debriefing and Rapid Cycle Deliberate Practice in Anaphylactic Shock Training on Nursing Students' Knowledge, Performance, Self-Confidence, and Satisfaction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, BETUL SAHIN KILINC, Lecturer in Nursing, MSc, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 171622998.600-294
Record Dates: First submitted 2026-01-21; First posted 2026-02-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Nursing Students; Nursing Education; Simulation Based Learning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): rapid cycle deliberate practice
  Interventions: Behavioral: rapid cycle deliberate practice
- Control group (Experimental): post-scenario debriefing
  Interventions: Behavioral: Post-scenario debriefing

INTERVENTIONS:
Behavioral: rapid cycle deliberate practice — Unlike traditional debriefing, feedback is provided by pausing the scenario within the simulation. Then the part of the script up to the pause point is repeated.
  Arms: Intervention Group
Behavioral: Post-scenario debriefing — Debriefing is performed at the end of the simulation scenario.
  Arms: Control group

SUMMARY:
This study aims to examine the effect of rapid cycle deliberate practice (RCDP) on nursing students' knowledge, performance, self-confidence, and satisfaction levels regarding anaphylactic shock management. Based on a randomized controlled study design, the study will compare third-year nursing students in terms of RCDP application with traditional analysis methods performed at the end of a scenario. Students, divided into intervention and control groups, will have their knowledge levels, simulation performance, self-confidence, and satisfaction assessed using various scales. The retention of learning and students' subjective learning experiences will also be included in the research. The outcome of this study will determine whether RCDP is an effective method for improving critical clinical decision-making and emergency management skills in nursing students.

ELIGIBILITY:
Inclusion Criteria:

* To agree to participate in the study:
* Being a 3rd year nursing student
* Not working as a nurse in a hospital or any healthcare facility

Exclusion Criteria:

* • Refusing to participate in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Nursing students' knowledge level regarding shock and anaphylactic shock: Knowledge Test Regarding Nursing Management in Anaphylactic Shock | before the intervention, on the day of the intervention, and 8 weeks after the intervention.
  Knowledge Test Regarding Nursing Management in Anaphylactic Shock The 'Knowledge Test Regarding Nursing Management in Anaphylactic Shock,' developed by researchers in line with the literature (Ren et al., 2022; Arslan, 2021; Wang et al., 2021; Karadakovan & Eti Aslan, 2017; Eti Aslan, 2017; Nair & Peate, 2018), will be administered as follows: a 'Pre-Test' before the training to determine the students' current knowledge level regarding shock and anaphylactic shock; a 'Post-Test' immediately following the simulation application after the training; and a '1st Retention Test' 8 weeks later to measure the retention of learning. The Knowledge Test consists of 25 multiple-choice questions with 5 options each, focusing on knowledge levels regarding shock and anaphylactic shock. This form has been finalized with necessary adjustments based on expert opinions. The maximum score on this test is 100 points, and the minimum is 0 points. A higher score indicates a higher level of knowledge.
Simulation Performance Checklist: Nursing Students' Performance Level Regarding Anaphylactic Shock | on the same day as the intervention and 8 weeks after the intervention
  Simulation Performance Checklist The 'Simulation Performance Checklist for Nursing Management in Anaphylactic Shock', created by researchers in line with the literature (Casale et al., 2023; Ren et al., 2022; Arslan, 2021; Dreborg and Him, 2021; Wang et al., 2021; Eti Aslan, 2017; Karadakovan, 2017), will be used to determine students' performance levels. A 'Post-Test' will be administered immediately after the simulation application, and a '1st Retention Test' will be administered after 8 weeks to measure the retention of learning. The checklist consists of 10 items, and each item is scored as "0 = Could not/Did not apply/No", "1 = Did/Applied/Yes". A minimum score of 0 and a maximum score of 10 can be obtained from the checklist. This form has been finalized after necessary adjustments were made in line with expert opinions.

SECONDARY OUTCOMES:
Student Satisfaction and Self-Confidence in Learning Scale: Self-confidence and satisfaction levels of nursing students | before the intervention and on the day of the intervention
  Student Satisfaction and Self-Confidence in Learning Scale The Student Satisfaction and Self-Confidence in Learning Scale was developed by Jeffries and Rizzolo (2006), and the Turkish adaptation, validity, and reliability study were conducted by Ünver et al. (2017). The scale consists of 12 items and has two sub-dimensions: student satisfaction (5 items) and self-confidence in learning (7 items). The scale is administered using a 5-point Likert scale (1=Strongly disagree - 5=Strongly agree). In the Turkish version, the Cronbach alpha coefficient was found to be between 0.77 and 0.85, showing that it is a valid and reliable measurement tool. A minimum score of 12 and a maximum score of 60 can be obtained from this scale. A score closer to 60 indicates positive results.
Debriefing Experience Scale | The simulation applications will be conducted on the same day.
  In this study, the Debriefing Experience Scale, developed by Reed (2012) and adapted into Turkish by Uslu et al. (2022), will be used as a data collection tool. The scale consists of 20 items and four sub-dimensions, and is a 5-point Likert type scale. The Cronbach's alpha coefficients of the Turkish form of the scale were determined as 0.948 for "Evaluation Experience" and 0.951 for "Importance of Item"; the test-retest reliability was ICC=0.999 (p<0.001). It was stated that the Turkish version is valid and reliable. A minimum score of 20 and a maximum score of 100 can be obtained from this scale. A score closer to 100 indicates positive results.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Ankara, Turkey (Türkiye)